CLINICAL TRIAL: NCT02657538
Title: Validation of Near-infrared Light Transillumination for Interproximal Enamel Caries Detection: A Clinical Controlled Trial
Brief Title: Validation of Near-infrared Light Transillumination for Interproximal Enamel Caries Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 110/13
Record Dates: First submitted 2016-01-05; First posted 2016-01-18 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Dental Caries
Keywords: Interproximal caries; Enamel caries; Caries detection; Caries diagnostics; Near-infrared light transillumination; DIAGNOcam
MeSH Terms: conditions — Dental Caries | interventions — Fluoridation; Observation; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Near infrared transillumination (Active Comparator): Near infrared transillumination is applied for initial enamel caries lesion detection.
  Interventions: Other: Non invasive caries treatment; Other: Invasive caries treatment; Device: Near-infrared light transillumination device (DIAGNOcam, KaVo, Biberach, Germany)
- Visual caries detection + BW (Active Comparator): visual caries detection + bite wing radiography (BW): considered as gold standard in caries diagnostics.
  Interventions: Other: Non invasive caries treatment; Other: Invasive caries treatment; Other: Visual examination and bitewing (BW) radiography

INTERVENTIONS:
Other: Non invasive caries treatment — If the active comparator does not detect cavitation, fluoride varnish is applied on the test surface.
  Other Names: Fluoridation
Other: Invasive caries treatment — If the active comparator does detect cavitation, a composite restauration is placed
  Other Names: Filling
Device: Near-infrared light transillumination device (DIAGNOcam, KaVo, Biberach, Germany)
  Arms: Near infrared transillumination
Other: Visual examination and bitewing (BW) radiography — established diagnostic methods
  Arms: Visual caries detection + BW

SUMMARY:
The aim of this study is to validate a near-infrared light transillumination device (DIAGNOcam, KaVo, Biberach, Germany) for interproximal enamel caries detection and compare it with the established diagnostic methods (visual examination and bitewing radiography). The aim is to avoid/reduce ionizing radiation for caries diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria:

* ASA-Status 1
* Complete permanent dentition
* Bitewing radiography already existing (< 4 months)
* Minimum of one cavitation-free approximal surface, symptomless, interproximal enamel or dentin caries lesion in the posterior teeth without restorations and/or sound tooth surface.

Exclusion Criteria:

* Children younger than 15 Years

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus W Neuhaus, PD, Principal Investigator — Department of Preventive, Restorative and Pediatric Dentistry, University of Bern

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: 35 participants with either initial caries and/or no carious lesion were included in this study.
  The participants had to be at least 14 years old, in good health (ASA-Status 1) and they had to give their informed consent.
Period: Overall Study
Arm/Group | All Study Participants
Started | 35
Received Near Infrared Transillumination | 35
Received Visual Caries Detection + Bite | 35
Completed | 31
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 27.5 [18 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Caries Extension According to Diagnocam Codes 0-4 (Intra- and Interrater-Reliability, Sensitivity and Specificity)
Description: The geometrical shape of caries lesions is displayed with the near infrared transillumination method. These shapes are classified as: code 0: no lesion visible; code 1: first visible signs in enamel; code 2: established, clear visible signs in enamel; code 3: clear visible in enamel and punctual contact with dentine; code 4: clearly visible and broad contact with dentine
  Intra- and Interrater-Reliability: Reliability indicates the overall consistency of a measurement. To have a high reliability means in this case, that the diagnostic-tool produces similar results under consistent conditions. The interrater-Reability assesses the degree of agreement between two different raters in their diagnostics on a specific test while the intrarater-Reliability assesses the degree of agreement of a single rater who did a diagnostic-test twice under the same testing conditions.
  Sensitivity and Specificity: Statistics are not done yet but will be updated when we calculated them
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: weighted Kappa
Units Other Than Participants: Teeth/ Leasons
Groups:
- Near Infrared Transillumination: Near infrared transillumination is applied for initial enamel caries lesion detection.
  Non invasive caries treatment: If the active comparator does not detect cavitation, fluoride varnish is applied on the test surface.
  Invasive caries treatment: If the active comparator does detect cavitation, a composite restauration is placed
  Near-infrared light transillumination device (DIAGNOcam, KaVo, Biberach, Germany)
Arm/Group | Near Infrared Transillumination | Visual Caries Detection + BW
Number analyzed (Participants) | 35 | 35
Number analyzed (Teeth/ Leasons) | 70 | 70
weighted Kappa
  Intra-rater agreement examiner 1 | 0.68 [0.39 to 0.70] | 0.87 [0.73 to 0.95]
  Intra-rater agreement examiner 2 | 0.62 [0.35 to 0.80] | 0.76 [0.58 to 0.86]
  Inter-rater agreement | 0.42 [0.13 to 0.42] | 0.60 [0.34 to 0.68]

2. Secondary Outcome: Lesion Activity
Description: active lesions: 1; inactive lesions: 0
Time Frame: One year
Population: The data were not collected and the Outcome will never be analyzed because of the study population. The participants are all low risk in the analysis of caries, with low amount of gingivitis and good oral hygiene what means that no progression/ change in caries activity will be detectable in any patient. So it doesn't make sense to analyze it.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Near Infrared Transillumination | Visual Caries Detection + BW
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes